CLINICAL TRIAL: NCT00544895
Title: Neonatal Estimation Of Brain Damage Risk And Identification of Neuroprotectants
Acronym: NEOBRAIN
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: European Commission (Other)
Responsible Party: Prof. Dr. med. Olaf Dammann, Perinatal Infectious Disease Epidemiology Unit - Medical School Hannover
Other Study IDs: LSHM-CT-2006-036534
Record Dates: First submitted 2007-10-12; First posted 2007-10-16 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2011-06

CONDITIONS: Brain Damage, Chronic
MeSH Terms: conditions — Brain Damage, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, urine
Oversight: Data Monitoring Committee: No

SUMMARY:
NEOBRAIN brings together small and medium sized enterprises (SMEs), industry and academic groups devoted to the diagnosis, management, and neuroprotection in newborns with perinatal brain damage. The focus of NEOBRAIN is to identify strategies prevention of brain damage mainly observed in preterm newborns. (Copy from www.neobrain.eu)

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 28 weeks

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Preterm newborns with a gestational age < 28wks
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2007-10; Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Brain white matter damage (WMD, defined by MRI ,US, EEG) | during stay in NICU and until discharge

SECONDARY OUTCOMES:
Developmental assessment | at 2 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Dammann, Study Director — Medical School Hannover
Locations (12):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Hôpital Robert Debré, Paris, France
- Germany (3):
  - Charité, Campus Virchow Klinikum, Berlin
  - Universität Duisburg-Essen, Essen
  - Hannover Medical School, Hanover
- Italy (2):
  - Fondazione I.R.C.C.S Ospedale Maggiore Policlinico MA.RE., Milan
  - Azienda Ospedaliera Universitaria Senese, Siena
- Wilhelmina Children's Hospital, Utrecht, Netherlands
- Sweden (3):
  - Perinatal Center, Gothenburg
  - University Hospital, Lund
  - Academic Children's Hospital, Uppsala
- Hôpital des Enfants, Geneva, Switzerland

REFERENCES:
- [Background] Dammann O, Cesario A, Hallen M. NEOBRAIN--an EU-funded project committed to protect the newborn brain. Neonatology. 2007;92(4):217-8. doi: 10.1159/000102967. Epub 2007 May 21. No abstract available. PMID 17992017